CLINICAL TRIAL: NCT05920902
Title: Arterial Spin Label Depicted Ischemic Stroke Cohort (ASLIS)
Acronym: ASLIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RJ_ASLIS
Record Dates: First submitted 2023-02-09; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-02

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemia stroke, arterial spin labeling, evaluation
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute ischemia stroke: Best medcine treatment. It including antiplatelet drugs, statins, hypotensive drugs, antidiabetics, neurotrophic drugs, butylphthalide, edaravone.
  Interventions: Other: routine therapy of acute ischemia stroke

INTERVENTIONS:
Other: routine therapy of acute ischemia stroke — Routine therapy of acute ischemia stroke based on the guidelines, which generally includes two parts: evaluation and medicine treatment. Evaluation includes peripheral blood test, radiologic examination, electrophysiological examination, ultrasonic examination. Medicine treatment includes drug therapy and rehabilitation.

SUMMARY:
Establish a clinical cohort of acute ischemic stroke patients and find the determinant of the prognosis.

DETAILED DESCRIPTION:
1. Enrollment: screening the candidates based on the inclusion and exclusion criteria, and sign the informed consent.
2. Baseline evaluation: evaluate baseline situation of enrolled candidates.
3. Inpatient view: view and evaluate enrolled candidates respectively at day 1, 3, 7 and 14 after stroke, and record the results.
4. Follow-up: view the candidates at 90 days and one year after stroke onset, and record the results.
5. Data analysis: analyze the results.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-90, no gender restrictions.
2. Onset of disease ≤7 days.
3. Meet either of the following two conditions:

   ① Transient ischemic attack (TIA)

   ② Ischemia stroke (IS) Note: Acute IS diagnosis criteria: sudden and persistent focal or widespread neurological dysfunction, excluding other non-vascular causes of brain dysfunction (such as brain infection, head injury, brain tumor, epilepsy, severe metabolic diseases, or degenerative neurological diseases), confirmed by image as new IS. TIA diagnosis criteria: sudden and reversible focal neurological or retinal ischemic deficit caused by a reversible ischemia, usually lasting less than 24 hours, with no evidence of new IS on imaging, and excluding other non-ischemic causes (such as brain infection, head injury, brain tumor, epilepsy, severe metabolic diseases, or degenerative neurological diseases).
4. Signed informed consent

Exclusion Criteria:

1. Clear cause of ischemic stroke other than atrial fibrillation.
2. Other ischemic strokes with a clear cause.
3. Presence of non-vascular intracranial disease.
4. Presence of severe systemic diseases.
5. Pregnancy or lactation.
6. Unable to tolerate or cooperate with MRI examination.
7. Unable to comply with follow-up due to geographical or other reasons.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Who sufferred acute ischemia stroke and be admitted to the ward of Ruijin Hospital, and meets the inclusion criteria, and does not meet the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progressively deterioration in acute phase | 7 days after ischemia stroke onset
  Number of participants whose SNOB (Standardised nursing observations for stroke) score at 7 days post ischemia stroke ≤ 2 points compared to baseline, and/or NIHSS score at 7 days post ischemia stroke ≥ 2 points compared to baseline are identified as progressively deterioration in acute phase.
Bad prognosis of acute ischemia stroke | 90 days after ischemia stroke onset
  Number of participants whose mRS (Modified rankin scale) score at 90 days after ischemia > 2 are identified as bad prognosis.

SECONDARY OUTCOMES:
Recurrent vascular episode | 1 year
  Including transient ischemia attack, intracranial hemorrhage, ischemia stroke
Recurrent artery stenosis | one year after stenting
  Degree of artery stenosis at one year after stenting > 50%
Unhealthy status | 1 year
  Any dimension in EQ-5D-3L (the generic three-level EuroQol five-dimensional questionnaire) score ≥ 2

CONTACTS AND LOCATIONS:
Overall Officials: Wei Jin, PhD. MD., Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Results of the research will be shared in the form of paper publishing. Other researchers who wants to know the details can contact with the PI.